CLINICAL TRIAL: NCT03708380
Title: Using a Geographically Targeted and Mixed Methods Approach to Improve Glycemic Control Among Black Men Identified as Having Previously Undiagnosed Diabetes and Prediabetes
Brief Title: Diabetes Prevention for Black Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-00826; R03DK120895 (Other Grant/Funding Number: NIH-NIDDK)
Record Dates: First submitted 2018-09-14; First posted 2018-10-17 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental): Community-based dietary intervention to Black and African American barbers identified as having previously undiagnosed diabetes and prediabetes
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Over a 60-day period, participants will receive healthy lunches that provide a hand-delivered healthy alterative to their current diets.

SUMMARY:
Geographic analyses of diabetes burden have found that poor glycemic control, high rates of diabetes-related hospital utilization, and a high prevalence of microvascular diabetic complications all cluster in the same neighborhoods.This proposed study seeks to identify Black barbers with undiagnosed diabetes or prediabetes using point-of-care HbA1c testing, perform qualitative interviews to identify health behaviors that may explain poor sugar control, and develop a workplace-based food intervention to promote primary prevention and test its effect on sugar control in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American men who work as barbers at Black-owned barbershops
* Barbershop clients.
* Workplace in neighborhood geographically identified as having higher diabetes burden
* No prior history of clinical diagnosis of diabetes
* Identified on initial and second point-of-care testing to have an HbA1c of 5.7 or greater

Exclusion Criteria:

* Individuals with a history of blood loss or blood disorder that would lead to incorrect results on point-of care HbA1c testing
* Individuals with a history of food allergies that requires specific dietary restrictions
* Individuals who are not English speaking
* Individuals who have a significant cognitive impairment that will be a barrier to communication, valid consent and participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Adherence to the intervention during the initial 60-day period when lunches are provided at no cost | 60 days
  Adherence will be calculated as the proportion of participants continuing to consume at least 80% of the lunch meals at the end of the initial intervention period when lunches will be provided at no cost.
Continuation with the dietary intervention after initial period when study participants may choose to pay for meals developed on their own | Until the end of the two year study period
  proportion of participants continue to purchase meals after the initial intervention period when individuals will be given the option to continue the intervention but paying for the lunch meals themselves.

SECONDARY OUTCOMES:
Photographic food and beverage diaries | Baseline
  Study participants will take photos of all food and beverages ingested over a 72-hourperiod to provide quantitative data on baseline dietary patterns
First Point-of-care Hemoglobin A1c (HbA1c) test | Baseline
  This first baseline point-of-care HbA1c test will be used as a reference.
Second Point-of-care HbA1C test | Baseline (3-6 months after first test)
  This second baseline point-of-care HbA1c test will be used to identify any changes in glycemic control that developed after initial diagnosis of diabetes or prediabetes by the first point-of-care test.
Third Point-of-care HbA1C test | Post treatment (3 months after the intervention)
  This post-treatment HbA1c test will be used to identify whether there was any short-term change in glycemic control after the dietary intervention
Fourth Point-of-Care HbA1c Test | Post-Treatment (6 to 12 months after the intervention)
  This post-treatment HbA1c test will be used to identify whether there was any longer-term change in glycemic control after the dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data. Requests should be directed to david.lee@nyumc.org. To gain access, data requestors will need to sign a data access agreement.